CLINICAL TRIAL: NCT01151709
Title: Assessment of Primary Care Providers' Knowledge and Beliefs Regarding Gout Management
Status: Completed | Type: Observational
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Leslie Harrold, Associate Professor of Medicine (UMMS), University of Massachusetts, Worcester
Other Study IDs: 13808
Record Dates: First submitted 2010-06-24; First posted 2010-06-28 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Gout
Keywords: Gout; Chronic condition management; Gout management
MeSH Terms: conditions — Gout

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- physicians: primary care practitioners, both family practice and internal medicine physicians from a random sample of providers nationwide

SUMMARY:
This is a questionnaire study aimed at learning about physicians' views on the treatment of Gout.

DETAILED DESCRIPTION:
We seek to assess the knowledge, beliefs and reported treatment practices of primary care physicians with regard to gout.

Specifically, we will:

* Assess the knowledge and beliefs with regard to acute and chronic gout management based on published treatment recommendations.
* Characterize the individuals who have knowledge deficits in terms of age, specialty, number of patients seen with gout, and practice setting.
* Assess the reported treatment practices of primary care physicians for the acute and chronic management of gout.

ELIGIBILITY:
Inclusion Criteria:

* practicing primary care practitioner, either in family medicine or internal medicine,
* must be 18 years of age or older

Exclusion Criteria:

* does not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care practitioners, both family practice and internal medicine physicians from a nationwide sample
Sampling Method: Probability Sample
Enrollment: 838 (Actual)
Dates: Start 2010-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Assess the knowledge and beliefs with regard to acute and chronic gout management based on published treatment recommendations. | 3 months
  Assess physicians' knowledge and beliefs with regard to acute and chronic gout management based on published treatment recommendations by means of questionnaire.
Characterize the individuals who have knowledge deficits in terms of age, specialty, number of patients seen with gout, and practice setting. | 3 months
  Characterize the individuals who have knowledge deficits in terms of age, specialty, number of patients seen with gout, and practice setting.
Assess the reported treatment practices of primary care physicians for the acute and chronic management of gout. | 3 months
  Assess the reported treatment practices of primary care physicians for the acute and chronic management of gout.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie R Harrold, MD, Principal Investigator — UMass Medical School
Locations (1):
- UMass Medical School, Worcester, Massachusetts, United States